CLINICAL TRIAL: NCT00264030
Title: Distal Protection Combined With PTCA in AMI Patients -- The DIPLOMAT Study.
Brief Title: Distal Protection Combined With PTCA in AMI Patients
Acronym: DIPLOMAT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Cordis US Corp. (Industry)
Responsible Party: Dr. Hans-Peter Stoll - Director Clinical Affairs, Cordis
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EC00-02
Record Dates: First submitted 2005-12-09; First posted 2005-12-12 (Estimated); Last update posted 2008-01-07 (Estimated); Status verified 2008-01

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Other): PTCA
  Interventions: Other: PTCA
- 2 (Other): PTCA with angioguard
  Interventions: Device: Angioguard distal protection device

INTERVENTIONS:
Device: Angioguard distal protection device — PTCA with the Angioguard distal protection device.
  Other Names: Cordis AngioGuard™ XP
  Arms: 2
Other: PTCA — PTCA
  Arms: 1

SUMMARY:
The primary objective is to evaluate if use of the AngioGuard™ XP improves myocardial reperfusion after PTCA as assessed by ST segment resolution at the end of PTCA.

DETAILED DESCRIPTION:
This is a prospective, randomized, multicenter trial. Patients will be randomized either to be treated by PTCA only or in combination with the An-gioGuard™ XP device. The patients will be followed for six-months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Acute myocardial infarction < 12 hours with ST segment elevation > 2 mm in at least 2 contiguous leads;
* Clinical indication of primary PTCA;
* De novo or restenotic lesions in native coronary vessel, single vessel treatment only;
* Target lesion stenosis is > 80% (by visual estimation).

Exclusion Criteria:

* Patient has unprotected left main coronary disease with > 50% stenosis in case left coronary artery is treated;
* Patient has an ostial target lesion;
* Killip class > 3.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2002-03; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Absolute ST segment resolution. | post-PTCA

SECONDARY OUTCOMES:
ST segment resolution (> 50% decrease). | pre- and post-PTCA
TIMI Frame Count | post PTCA
Composite endpoint of slow flow, no reflow or distal embolization. | at anytime
Regional wall motion index by echocardiography. | discharge and 6 month follow-up
Clinical success evaluation; qualitative evaluation of device and delivery system characteristics. | post-procedure
Cardiac function assessed by echocardiography. | before discharge and at 6 month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Thierry LEFEVRE, MD, Principal Investigator — Hopital Tarnier-Cochin
Locations (1):
- Institut Cardiovasculaire Paris Sud, Massy, France